CLINICAL TRIAL: NCT07076953
Title: The Effect of Cherry Pitted Massage on Primiparous Pregnant Women During Labor on Postpartum Lactation Onset Symptoms and Insufficient Milk Perception: A Randomized Controlled Trial
Brief Title: Cherry Seed Massage Lactation and Milk Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Hafizenur Karaduman, Graduate Student, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KaratayU-SBF-HK-01
Record Dates: First submitted 2025-07-08; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Breast-feeding; Massage Effect; Primiparity
Keywords: Labor; Lactation; Cherry pit massage; Perception of insufficient milk; Manual massage; Breastfeeding; Midwife support
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: There is a manual massage group, a cherry seed massage group , a control group. The Effect of Cherry Pitted Massage on Primiparous Pregnant Women During Labor on Postpartum Lactation Onset Symptoms and Insufficient Milk Perception
Who Masked: Outcomes Assessor
Masking Description: The statistician was blinded in the study. The researcher blinding was not done because he was the implementer. In order to prevent bias in the evaluation of the data; groups A, B and C were coded by an independent academician other than the researcher and the data were analyzed by an independent statistician. After the analysis and interpretation of the data were completed, the codes of the intervention and control groups of the study were revealed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hand Massage Group (Active Comparator): Data collection in the study was conducted in a planned and structured manner, starting from the third stage of labor. Participants in the intervention groups (manual massage and cherry pit massage) received two 15-minute massages, one in the first hour and one in the second hour postpartum, after the third stage of labor was completed. During the treatment, the mother's position was adjusted appropriately, with privacy and comfort prioritized, and intervention was interrupted in the event of pain or discomfort. During the data collection process, signs of the onset of lactation (breast fullness, milk leakage, tingling, etc.) were observed within the first 24 hours after birth for all three groups (manual massage, cherry pit massage, and the control group), and mothers' perception of insufficient milk supply was assessed using structured questionnaires and scales.
  Interventions: Other: Manual Breast Massage
- Cherry Pit Massage Group (Active Comparator): Data collection in the study was conducted in a planned and structured manner, starting from the third stage of labor. Participants in the intervention groups (manual massage and cherry pit massage) received two 15-minute massages, one in the first hour and one in the second hour postpartum, after the third stage of labor was completed. During the treatment, the mother's position was adjusted appropriately, with privacy and comfort prioritized, and intervention was interrupted in the event of pain or discomfort. During the data collection process, signs of the onset of lactation (breast fullness, milk leakage, tingling, etc.) were observed within the first 24 hours after birth for all three groups (manual massage, cherry pit massage, and the control group), and mothers' perception of insufficient milk supply was assessed using structured questionnaires and scales.
  Interventions: Other: Cherry Seed Massage Group
- Control Group (No Intervention): No intervention other than routine care was applied to the control group of the study, and research data were collected at simultaneous intervals with the intervention groups.

INTERVENTIONS:
Other: Cherry Seed Massage Group — In the third stage of labor, a cherry pit massage was applied for 15 minutes in the first and second hours. Cherry pits were added to a silk bag to prevent damage to the skin during the massage. The massage application steps were applied as indicated in the hand massage
  Arms: Cherry Pit Massage Group
Other: Manual Breast Massage — Manual massage was applied for 15 minutes during the third stage of labor, first and second hour.Manual breast massage steps; Step 1: The breast tissue under and near the armpit is compressed and released like a water pump.
  Step 2: Pressure is applied to the breast tissue. Step 3: The breasts are massaged using the fingers and pressed with small circular movements. It is moved clockwise and counterclockwise around the breast and towards the areola with light touches.
  Step 4: Both hands are placed under the breast; the breast is moved up and down, left and right, forward and backward.
  Step 5: One hand is placed under the breast and the other hand is on the breast; the hands are moved in the opposite direction and a rolling motion is applied to the breast.
  Arms: Hand Massage Group

SUMMARY:
The perception of insufficient milk is quite common in mothers during the postpartum period. Especially mothers who have given birth for the first time tend to external factors more due to lack of experience. Studies mention many nonpharmacological methods to prevent this. Some of these are hypnobreastfeeding, hot application, breast massage, aromatherapy. There are many studies on breast massage to increase milk to date. However, no study with cherry seed has been identified. By eliminating the deficiency in the literature and proving the effect of cherry seed breast massage on insufficient milk perception and lactation start-up symptoms, it will be ensured that breastfeeding is not terminated early, and this research is needed considering the perspective of improving mother and baby health by breastfeeding for the first 6 months. The study will be conducted in a single-blind randomized control design. The study will be conducted in Konya Medova Hospital. A total of 54 puerpera will be included in the study, including the cherry seed massage intervention group (18), the hand massage intervention group (18), and the control group (18). The study data will be collected using the Introductory Information Form, the Insufficient Milk Perception Scale, and the Visual Analog Scale (Vas) to Evaluate Mothers' Lactation Initiation Symptoms. The intervention group data will be collected in the first five minutes, 30 minutes, 1 hour, and 2 hours after birth. SPSS 23 (IBM, Inc., Armonk, NY, USA) program will be used in the analysis and evaluation of the data. The results obtained will be tested at a significance level of p<0.05 and two-way.

DETAILED DESCRIPTION:
Breast milk is the ideal food source, containing all the nutrients that meet all the needs of the newborn and supporting immunity with its bioactive content . The World Health Organization (WHO), the United Nations Children's Fund (UNICEF), the American Academy of Pediatrics (APA), and the Ministry of Health (MoH) recommend that babies should be exclusively breastfed for the first six months, and that breastfeeding should continue with complementary foods until the age of two. Breast milk meets all of the energy and nutritional needs of the baby in the first six months, more than half after the sixth month, and one-third until the second year.

Data from the Turkey Demographic Health Survey (TDHS) show that breastfeeding is very common in Turkey, with 98% of infants breastfed in the two years prior to the survey. However, 41% of infants under 6 months of age in Turkey are exclusively breastfed, and the median duration of exclusive breastfeeding is 1.8 months . Many women, despite being able to produce enough milk to meet their baby's milk needs, worry that it's not enough. This is cited as one of the most common reasons for prematurely ending breastfeeding or supplementing with formula . The perception of insufficient milk stems from mothers' concerns that the quality and quantity of milk are insufficient for their babies, and their belief that their babies are not getting enough. The "perception of insufficient milk supply," which cannot be expressed with objective data and is simply assumed to be "there," is one of the leading reasons for not continuing breastfeeding . Furthermore, while more than 50% of breastfeeding mothers perceive their milk supply as insufficient, it is reported that only 5% actually experience physiological milk insufficiency . Therefore, midwives are expected to provide breastfeeding counseling in the postpartum period and contribute to the continuation of breastfeeding by reducing mothers' perception of insufficient milk supply through accurate information and psychosocial support. Harting et al. (2025) state that midwives reinforce mothers' confidence in the breastfeeding process and play an important role in encouraging breastfeeding through practices such as breastfeeding initiation, skin-to-skin contact, and breastfeeding counseling. Breast massage applied within this scope has been reported to support the early onset of lactation and is effective in reducing mothers' perception of insufficient milk supply. The literature reports that oketani massage increases breastfeeding success and reduces the time to breastfeeding initiation and breast massage combined with acupuncture stimulation increases breast milk production . It has also been reported that breast massage combined with milk expression increases breast milk production by 92% and the average daily milk supply by 48%, while reducing pumping duration and frequency .

There are also various scientific studies on the materials used in breast massage treatments in the delivery room. A therapy device called BERES, designed to massage and heat the breasts, has been reported to increase breast milk production from 20 ml before use to 27.3 ml after use . The Lactamo breast massage device, which combines heating/cooling and compression, has been reported to be beneficial for pain, congestion, and milk production problems . The Gua Sha massage technique, commonly used in traditional Chinese medicine by scraping the skin with smooth stones like jade, has been reported to help increase lymphatic drainage and relieve breast congestion . Products like Lansinoh Therapearl and Mumasil Reusable Warm and Cool Breast Packs are disc-shaped gel packs designed for this purpose. These packs are warmed before breastfeeding to encourage milk flow and cooled after breastfeeding to reduce pain and swelling . Similarly, cherry pit sachets, used as natural heat traps and massage tools, are thought to stimulate milk ducts when applied to breast tissue, facilitating the onset of lactation.

This study aims to evaluate the effects of massage with cherry pit sac applied to primiparous pregnant women during labor on physiological signs of postpartum lactation and mothers' perception of insufficient milk supply. While the literature indicates the positive contributions of breast massage and hot and cold applications to the lactation process, studies directly examining the effect of massage applied during labor on postpartum milk production are limited. Furthermore, the potential benefits of using cherry pit sac, a natural, accessible, and noninvasive method, in this process have not been adequately documented in the literature. Cherry pit sacs, with their natural structure that allows them to retain heat for extended periods and distribute evenly across the body when applied, have the potential to be an ideal material for massage applications. Furthermore, it is anticipated that this method may reduce the perception of insufficient milk supply, a common complaint among mothers, and support the continuity of breastfeeding. In this respect, the study has the potential to make an ecological and cost-effective contribution to postpartum care practices. The lack of scientific data in the literature on the use of cherry pit as a breastfeeding support material constitutes both the innovative aspect and the scientifically original value of this study.

Hypotheses

H1. Massage with cherry pits in primiparous pregnant women during labor accelerates the onset of postpartum lactation symptoms.

H2. Massage with cherry pits in primiparous pregnant women during labor reduces the perception of insufficient postpartum milk supply.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years of age,
* 37-42 weeks of pregnancy,
* Primiparous,
* Able to read and write Turkish,
* Volunteer women were included in the study

Exclusion Criteria:

* Women who have a risky pregnancy (such as IVF pregnancy, multiple pregnancy, preeclampsia),
* Women who smoke or use alcohol,
* Women who have a physiological or anatomical obstacle that may prevent lactation,
* Women who have infectious diseases such as HIV, Hepatitis B, Hepatitis C, which are known to be transmitted through breast milk, were excluded.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 54 (Actual)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Insufficient Milk Perception Scale | Between 5-35 minutes after birth,in the first hour after birth, in the second hour after birth, for fifteen minutes
  The Turkish validity and reliability study was conducted by Gökçeoğlu and Küçükoğlu (2014). The scale consists of 6 questions. The first question, which asks whether the mother perceives her milk supply as sufficient, is answered with a "yes" or "no" question. The other 5 questions measure the perception of insufficient milk supply and are scored from 0 to 10. The scale is scored from 0 to 50. Cronbach's alpha was determined as 0.81 in the original scale and was found to be 0.82 in the Turkish validity and reliability study. In this study, Cronbach's alpha values were found to be highly reliable at 0.757 for the pretest, highly reliable at 0.881 for the third stage of labor, highly reliable at 0.91 for the first hour, and highly reliable at 0.931 for the second hour.

SECONDARY OUTCOMES:
Lactation Evaluation Form | Between 5-35 minutes after birth,in the first hour after birth, in the second hour after birth, for fifteen minutes
  The "Lactation Assessment" section of the Lactation, Infant Suckling Behavior, and First Breastfeeding Assessment Form, developed by Tatarlar and Tokat (2015) and used in their master's thesis, was used. The form assesses breast fullness, milk letdown, and post-breastfeeding status. In the study, the form was evaluated as a categorical variable and analyzed using numbers and percentages. The form was completed by the researcher using physical examination and observation methods.

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay Üniversitesi, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No